CLINICAL TRIAL: NCT03099863
Title: Cytoscopic Antibiotic Irrigant to Reduce Postoperative Urinary Infection: A Randomized Controlled Study
Brief Title: Cytoscopic Antibiotic Irrigant to Reduce Postoperative Urinary Tract Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Mangel, Physician, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB15-00769
Record Dates: First submitted 2017-03-23; First posted 2017-04-04 (Actual); Results first posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cystoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (Placebo Comparator): Standard cystoscopy with normal saline solution.
  Interventions: Procedure: Cystoscopy; Drug: Cystoscopic Fluid/Placebo
- Neosporin G. U. Irrigant (Active Comparator): Standard cystoscopy with normal saline solution containing Neosporin® G.U. at a 1mL/1000mL concentration.
  Interventions: Drug: Cystoscopic Fluid containing Neosporin G. U. Irrigant; Procedure: Cystoscopy

INTERVENTIONS:
Drug: Cystoscopic Fluid containing Neosporin G. U. Irrigant — Normal saline cystoscopic fluid containing Neosporin G. U. Irrigant 1mL/1000mL
  Arms: Neosporin G. U. Irrigant
Procedure: Cystoscopy — Diagnostic cystoscopy performed during pelvic floor surgery
Drug: Cystoscopic Fluid/Placebo — Normal saline cystoscopic fluid
  Arms: Standard Care

SUMMARY:
Postoperative urinary tract infections (UTIs) affect 20-30% of patients undergoing elective gynecologic surgery and have a significant socioeconomic impact and cost. Preoperative antibiotics, sterile operating techniques, postoperative antibiotic and non-antibiotic medical therapies have been utilized to attempt to decrease this rate with little improvement. Utilization of an intraoperative antibiotic cystoscopic irrigant may decrease postoperative UTIs. The investigators have designed a prospective randomized controlled study to evaluate the effectiveness of an antibiotic cystoscopic fluid in preventing postoperative urinary tract infections in women undergoing elective pelvic floor surgery with cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult women at least 18 years of age
* Elective Female Pelvic Medicine and Reconstructive Surgery or Gynecologic Minimally Invasive surgeries including hysterectomy, suburethral sling, and pelvic organ prolapse repair that require cystoscopy.

Exclusion Criteria:

* Surgeries that include: intradetrusor Botox, vaginal mesh excision, and fistula repair
* Pregnancy
* History of nephrolithiasis
* Allergy to study medications
* Congenital urogenital anomaly
* Neurogenic bladder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Neosporin G. U. Irrigant
Started | 121 | 121
Completed | 111 | 105
Not Completed | 10 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Neosporin G. U. Irrigant | Total
Number analyzed (Participants) | 111 | 105 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (1.0) | 51.2 (1.1) | 51.6 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 105 | 216
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Population: All participants were analyzed
  participants
    White | 62 | 60 | 122
    African American | 34 | 33 | 67
    Latina | 12 | 12 | 24
    Other | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 111 | 105 | 216
Surgery Type (patients could have more than 1 procedure) [Number; unit: participants]
  Vaginal Hysterectomy | 79 | 68 | 147
  Uterosacral ligament suspension | 14 | 16 | 30
  Vaginal native tissue repair | 19 | 14 | 33
  Midurethral sling | 62 | 46 | 108
  Laparoscopic surgery | 41 | 45 | 86

OUTCOME MEASURES:

1. Primary Outcome: Urinary Tract Infection
Description: Urinary tract infection defined as positive urinalysis, urine culture, and/or positive lower urinary tract symptoms requiring antibiotic treatment.
Time Frame: 4 weeks
Measure: Number (80% Confidence Interval); unit: UTI
Arm/Group | Standard Care | Neosporin G. U. Irrigant
Number analyzed (Participants) | 111 | 105
UTI | 11 [4 to 16] | 12 [5 to 18]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Standard Care | Neosporin G. U. Irrigant
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/105
Other Adverse Events (participants affected / at risk) | 0/111 | 0/105

LIMITATIONS AND CAVEATS:
Our primary limitation is the failure to reach statistical power based on the lower than expected incidence of UTI. Additionally, our patient cohort had a wide variation in surgical approach and techniques, which have different UTI risks at baseline. The total cohort is underpowered to identify differences in any one procedure type, such as vaginal reconstruction or mid-urethral slings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT03099863/Prot_SAP_000.pdf